CLINICAL TRIAL: NCT05935228
Title: Development and Evaluation of an Algorithm for Vascular Access Management - ALCOV Pilot Study
Brief Title: Development and Evaluation of an Algorithm for Vascular Access Management
Acronym: ALCOV
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, SLOSSE Come, Principal Investigateur, Central Hospital, Nancy, France
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2023-A00223-42
Record Dates: First submitted 2023-05-09; First posted 2023-07-07 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Peripheral Venous Access
Keywords: Difficult Intravenous Access (DIVA); Difficult Intravenous Access Scale (A-DIVA Scale); Algorithm; Peripheral venous catheter; Decision-making tree

STUDY DESIGN:
Intervention Model Description: This is a mixed (quantitative and qualitative), multicentre, non-randomised, quasi-experimental, before-and-after, open, cross-sectional study, with control and experimental groups and comprising three phases. This division into three data collection phases allows detailed analysis of the targeted care procedure and avoids errors of assessment of the impact of the different tools introduced in the interventional phase (the vascular access difficulty score [VAD] in phase 2, then the algorithm [composed of the VAD score and the graded decision tree for management] in phase 3).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- The control group (Other): The control group will consist of patients included in phase 1. These are the patients from the "before" phase, i.e. before the implementation of the Difficult Intravenous Access Scale.
  Interventions: Other: Implementation of the A-DIVA Scale
- The experimental group (Experimental): The experimental group will consist of the patients included in phase 3. These are the patients from the "after" phases i.e after the implementation of the algorithm.
  Interventions: Other: Implementation of the algorithm composed of the A-DIVA Scale and the new decision-making tree (the A-DIVA Tool) in the centers

INTERVENTIONS:
Other: Implementation of the A-DIVA Scale — Phase 2 aims to evaluate the impact of the implementation of the A-DIVA Scale (classification score for difficult intravenous access) on practitioners' approaches to the peripheral venous catheter placement. It consists of a systematic collection of peripheral venous catheter placement practices for quantitative data and a questionnaire of professionals' opinions on the use of the A-DIVA scale for qualitative data. The main objective of this phase is to recognize the potential appearance of changes in practices through the implementation of a tool for evaluating vascular access difficulties
  Arms: The control group
Other: Implementation of the algorithm composed of the A-DIVA Scale and the new decision-making tree (the A-DIVA Tool) in the centers — The main objective of this phase is to evaluate the impact of the algorithm on the quality of peripheral venous catheter placement.
  • Systematic collection of judgment criteria and socio-demographic and clinical characteristics of patients. Description of the care strategy implemented. Systematic collection of the A-DIVA Scale with identification of the patient's risk group, systematic rating of pain and evaluation of overall comfort.
  Arms: The experimental group

SUMMARY:
Two billion catheters are placed annually worldwide. Of all the people requiring vascular access, nearly a quarter have Difficult Intravenous access (DIVA), a source of multiple punctures. The increased risk of haematomas, haemorrhages, infection, pain and associated trauma is responsible for increased human costs and economic impact.

To limit the risks posed by the DIVA, practitioners have solutions such as the per-bone line, other types of lines, and placement of peripheral venous catheter with ultrasound or transluminescence. However, these solutions are not always applicable, depending on the care situation (non-substitutable venous access, fragile patient, etc.) or on the technical platform (available personnel and training, configuration of the premises, available equipment). Moreover, these actions are often taken after failures, in a non-anticipated and non-consensual manner.

In order to assess the risk of DIVA, F.Van Loon et al developed in 2016, and then modified in 2018, a DIVA Scale (the A-DIVA Scale) which allows a rapid scoring upstream of peripheral venous catheter placement to classify patients according to the risk of DIVA.

Composed of five items (non-palpable and non-visible vein, diameter < 3mm, history of DIVA, operator experience) worth one point each, the score allows three categories to be established: "low risk", "moderate risk", "high risk". The study showed that the proportion of first puncture failures increased with the risk of the patients (defined according to the categorized score).

The use of a tool such as the A-DIVA Scale is of interest if it allows the definition of actions to be taken in relation to the risk it identifies. In view of this, it appears essential to optimize the management of peripheral venous catheters, particularly for patients with DIVAs. The aim of this study is to develop a graduate and specific response to the issue of multiple punctures. Our project is to create and evaluate a specific algorithm, consisting of a risk assessment (the A-DIVA Scale) and a co-construct decision-making tree (the A-DIVA Tool). Built on the basis of objective clinical data collection and adapted to the possibilities and competencies, this new tool would bring real benefits to the patient in terms of safety (reduction of risks) and comfort (reduction of pain and duration of management), as well as a medico-economic benefit for the institutions. To date, such an algorithm does not exist and its beneficial effects have not been evaluated.

DETAILED DESCRIPTION:
This is a mixed (quantitative and qualitative), multicentre, non-randomised, quasi-experimental, before-and-after, open, cross-sectional study, with control and experimental groups and comprising three phases. This division into three data collection phases allows detailed analysis of the targeted care procedure and avoids errors of assessment of the impact of the different tools introduced in the interventional phase (the A-DIVA Scale in phase 2, then the algorithm [composed of the A-DIVA Scale and the new decision-making tree (A-DIVA Tool] in phase 3).

Phase 1 (observational: 4 months): Description of the inclusion centers and collection of pre-intervention data.

This phase will provide information on the actual practices and organization in the inclusion centers. The main objective of this phase is to provide a detailed description of existing practices for peripheral venous catheter placement in the inclusion centers.

It consists of individual semi-directive explanatory interviews with healthcare professionals in the inclusion centers, and a collection of judgment criteria (excluding the feelings of patients and caregivers concerning the implementation of the DIVA score and the catheter placement algorithm). Collection of socio-demographic and clinical characteristics of patients and description of the care strategy implemented.

Phase 2 (interventional: 4 months - implementation of the A-DIVA Scale alone): Collection of data related to the isolated implementation of a systematic scoring of the A-DIVA score.

Phase 2 aims to evaluate the impact of the implementation of the A-DIVA Scale (classification score for DIVA) on practitioners' approaches to the peripheral venous catheter placement. It consists of a systematic collection of peripheral venous catheter placement practices for quantitative data and a questionnaire on the opinions of professionals on the use of the A-DIVA Scale for qualitative data. The main objective of this phase is to recognize the potential appearance of changes in practices through the implementation of a score for evaluating DIVA (compared with the initial practices clarified in phase 1).

Compared to phase 1: addition of systematic collection of the A-DIVA Scale with identification of the patient's risk group, systematic rating of pain and assessment of overall comfort.

Interphase: (8 months) Co-construction of the decision-making tree (the A-DIVA Tool).The interphase will allow to analyze the data collected in phase 1 and phase 2 and to develop the algorithm (composed by the A-DIVA Scale and the new A-DIVA Tool).

1. Organization of a working group (including the investigator and volunteer caregivers): The data acquired in phase 1 and 2 will be described and presented to the professionals of each center in order to provide a basis for co-constructing the decision-making tree during the work groups.
2. Validation of the algorithm according to the A-DIVA Scale based on literature data, research hypotheses and working group data. Presentation of the model to the care teams, validation of its acceptability and feasibility.

Phase 3 (interventional: 4 months - use of the algorithm composed of the A-DIVA Scale and the Co-constructed decision-making tree [The A-DIVA Tool]): Implementation and evaluation of the algorithm in the centers. The main objective of this phase is to evaluate the impact of the algorithm on the quality of peripheral venous catheter placement.

* Systematic collection of judgment criteria and socio-demographic and clinical characteristics of patients. Description of the care strategy implemented (algorithm). Systematic collection of the A-DIVA Scale with identification of the patient's risk group, systematic rating of pain and evaluation of overall comfort.
* In relation to phase 2: implementation of the algorithm and collection of data to evaluate the implementation of the algorithm (e.g., frequency of use, optimal implementation (yes/no))

Post processing - valorization (10 months): Data analysis and scientific production:

The post-processing will allow the analysis of all the data (phase 3 versus phase 1 in particular), the production of reports and scientific articles and the writing of the final report of the ALCOV study.

* Analysis of the satisfaction questionnaire (proposed to caregivers at the end of the study) to complete the evaluation of the implementation of the algorithm.
* Description of the data (global and phase-by-phase) and analysis of the data to answer the formulated objectives, coding of the data from the interviews and satisfaction questionnaires, production of reports and scientific articles.

Representativeness of the sample:

- Throughout the collection process (phase 1,2 and 3) the representativeness of the sample will be assessed. The data collected for this purpose will be, for each patient who has received a peripheral venous line and who meets the inclusion criteria: Included: yes/no, if no: reason.

ELIGIBILITY:
Inclusion Criteria:

* Patient inclusion criteria: adult patients, initially requiring at least one peripheral venous catheter (PVC), having given their consent for the study.
* Inclusion criteria for healthcare professionals: Nurses, specialized nurses (IADE) and physicians attached to the department.

Exclusion Criteria:

Patient exclusion criteria :

* Minor patients
* Patients under curators or guardianship
* Patients who are non-communicative or unable to give consent
* Patients not requiring a peripheral venous catheter, polytrauma patients and patients in shock (septic, hemorrhagic, cardiogenic, spinal, specific to certain centers and equipped upstream)
* Patients who already have catheters on arrival.

Exclusion criteria for healthcare professionals: any professional not attached to the department and other professional categories.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 794 (Estimated)
Dates: Start 2023-12-05 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-09 (Estimated)

PRIMARY OUTCOMES:
1. Number of venipunctures performed per patient after implementation of the algorithm | 20 months
  Number of punctures performed per patient after implementation of the algorithm (collection according to a data grid filled in by the operator after the care).

SECONDARY OUTCOMES:
2. Number of participants who approve the co-constructed algorithm. | 8 months
  Co-construct a catheter placement algorithm based on the venous access difficulty score
3. Acceptability and feasibility of using the VAD score in isolation and the score in conjunction with the catheter placement algorithm | 4 months
  To meet this objective, caregivers' appreciation, use and feelings regarding the vascular access difficulties score and algorithm will be measured using a 23-item questionnaire scored on a 4-point Likert scale ("strongly disagree", "disagree", "agree", "strongly agree"). This questionnaire will also measure the effect of the vascular access difficulties score and the algorithm on practices.
Patient pain score measured immediately after vascular puncture (phase of potential acute pain during catheter insertion) using a self-assessment tool (numerical scale ranging from 0: no pain; 10: maximum pain) | 8 months and 16 months
  Describe how patients feel in terms of pain during care and overall comfort before and after the implementation of a catheter placement algorithm
5. Number of venipunctures performed per patient after implementation of the venous access difficulty score | 8 months
  Evaluate the effect of implementing the venous access difficulty score on the average number of venipunctures per patient
Insertion technique used for catheter placement | 8 months ans 16 months
  Assessing operators' professional practices
Number of operators required for catheter insertion | 8 months ans 16 months
  Assessing operators' professional practices
Frequency of second-line referral to another practitioner | 8 months ans 16 months
  Assessing operators' professional practices
Puncture result: success/failure | 8 months ans 16 months
  Assessing operators' professional practices
Care strategies implemented in the event of difficulties encountered when inserting peripheral venous lines collected by the operator at the end of care. | 8 months ans 16 months
  Strategies implemented in the event of difficulties will be measured using a multi-modality question (several answers possible): Call another practitioner, use an alternative insertion technique, choose another type of venous line, give up

CONTACTS AND LOCATIONS:
Overall Officials: Côme SLOSSE, Principal Investigator — Center Hospital Nancy
Locations (1):
- Center Hospital Nancy, Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rickard CM, Marsh N, Webster J, Runnegar N, Larsen E, McGrail MR, Fullerton F, Bettington E, Whitty JA, Choudhury MA, Tuffaha H, Corley A, McMillan DJ, Fraser JF, Marshall AP, Playford EG. Dressings and securements for the prevention of peripheral intravenous catheter failure in adults (SAVE): a pragmatic, randomised controlled, superiority trial. Lancet. 2018 Aug 4;392(10145):419-430. doi: 10.1016/S0140-6736(18)31380-1. Epub 2018 Jul 26. PMID 30057103
- [Background] van Loon FHJ, Buise MP, Claassen JJF, Dierick-van Daele ATM, Bouwman ARA. Comparison of ultrasound guidance with palpation and direct visualisation for peripheral vein cannulation in adult patients: a systematic review and meta-analysis. Br J Anaesth. 2018 Aug;121(2):358-366. doi: 10.1016/j.bja.2018.04.047. Epub 2018 Jul 2. PMID 30032874
- [Background] Bauman M, Braude D, Crandall C. Ultrasound-guidance vs. standard technique in difficult vascular access patients by ED technicians. Am J Emerg Med. 2009 Feb;27(2):135-40. doi: 10.1016/j.ajem.2008.02.005. PMID 19371518
- [Background] Adhikari S, Blaivas M, Morrison D, Lander L. Comparison of infection rates among ultrasound-guided versus traditionally placed peripheral intravenous lines. J Ultrasound Med. 2010 May;29(5):741-7. doi: 10.7863/jum.2010.29.5.741. PMID 20427786
- [Background] Bjorkander M, Bentzer P, Schott U, Broman ME, Kander T. Mechanical complications of central venous catheter insertions: A retrospective multicenter study of incidence and risks. Acta Anaesthesiol Scand. 2019 Jan;63(1):61-68. doi: 10.1111/aas.13214. Epub 2018 Jul 11. PMID 29992634
- [Background] Marsh N, Larsen EN, Takashima M, Kleidon T, Keogh S, Ullman AJ, Mihala G, Chopra V, Rickard CM. Peripheral intravenous catheter failure: A secondary analysis of risks from 11,830 catheters. Int J Nurs Stud. 2021 Dec;124:104095. doi: 10.1016/j.ijnurstu.2021.104095. Epub 2021 Sep 26. PMID 34689013
- [Background] Liu YT, Alsaawi A, Bjornsson HM. Ultrasound-guided peripheral venous access: a systematic review of randomized-controlled trials. Eur J Emerg Med. 2014 Feb;21(1):18-23. doi: 10.1097/MEJ.0b013e328363bebc. PMID 23880981
- [Background] Bouaziz H, Zetlaoui PJ, Pierre S, Desruennes E, Fritsch N, Jochum D, Lapostolle F, Pirotte T, Villiers S. Guidelines on the use of ultrasound guidance for vascular access. Anaesth Crit Care Pain Med. 2015 Feb;34(1):65-9. doi: 10.1016/j.accpm.2015.01.004. Epub 2015 Mar 5. PMID 25829319
- [Background] Cai EZ, Sankaran K, Tan M, Chan YH, Lim TC. Pen Torch Transillumination: Difficult Venepuncture Made Easy. World J Surg. 2017 Sep;41(9):2401-2408. doi: 10.1007/s00268-017-4050-3. PMID 28484817
- [Background] Adams DZ, Little A, Vinsant C, Khandelwal S. The Midline Catheter: A Clinical Review. J Emerg Med. 2016 Sep;51(3):252-8. doi: 10.1016/j.jemermed.2016.05.029. Epub 2016 Jul 5. PMID 27397766
- [Background] Lockwood J, Desai N. Central venous access. Br J Hosp Med (Lond). 2019 Aug 2;80(8):C114-C119. doi: 10.12968/hmed.2019.80.8.C114. PMID 31437056
- [Background] Vinan-Vega MN, Rahman MR, Thompson J, Ruppert MD, Patel RJ, Ismail A, Mousa S, Payne JD. Air embolism following peripheral intravenous access. Proc (Bayl Univ Med Cent). 2019 Jun 3;32(3):433-434. doi: 10.1080/08998280.2019.1609154. eCollection 2019 Jul. PMID 31384213
- [Background] Loon FHJV, Puijn LAPM, Houterman S, Bouwman ARA. Development of the A-DIVA Scale: A Clinical Predictive Scale to Identify Difficult Intravenous Access in Adult Patients Based on Clinical Observations. Medicine (Baltimore). 2016 Apr;95(16):e3428. doi: 10.1097/MD.0000000000003428. PMID 27100437
- [Background] van Loon FHJ, van Hooff LWE, de Boer HD, Koopman SSHA, Buise MP, Korsten HHM, Dierick-van Daele ATM, Bouwman ARA. The Modified A-DIVA Scale as a Predictive Tool for Prospective Identification of Adult Patients at Risk of a Difficult Intravenous Access: A Multicenter Validation Study. J Clin Med. 2019 Jan 26;8(2):144. doi: 10.3390/jcm8020144. PMID 30691137
- [Background] Bahl A, Johnson S, Alsbrooks K, Mares A, Gala S, Hoerauf K. Defining difficult intravenous access (DIVA): A systematic review. J Vasc Access. 2021 Nov 17;24(5):904 - 910. doi: 10.1177/11297298211059648. Print 2023 Sep. PMID 34789023
- [Background] Civetta G, Cortesi S, Mancardi M, De Pirro A, Vischio M, Mazzocchi M, Scudeller L, Bottazzi A, Iotti GA, Palo A. EA-DIVA score (Enhanced Adult DIVA score): A new scale to predict difficult preoperative venous cannulation in adult surgical patients. J Vasc Access. 2019 May;20(3):281-289. doi: 10.1177/1129729818804994. Epub 2018 Oct 16. PMID 30324841
- [Background] Girotto C, Arpone M, Frigo AC, Micheletto M, Mazza A, Da Dalt L, Bressan S. External validation of the DIVA and DIVA3 clinical predictive rules to identify difficult intravenous access in paediatric patients. Emerg Med J. 2020 Dec;37(12):762-767. doi: 10.1136/emermed-2020-209658. Epub 2020 Oct 20. PMID 33082150
- [Background] Santos-Costa P, Sousa LB, van Loon FHJ, Salgueiro-Oliveira A, Parreira P, Vieira M, Graveto J. Translation and Validation of the Modified A-DIVA Scale to European Portuguese: Difficult Intravenous Access Scale for Adult Patients. Int J Environ Res Public Health. 2020 Oct 17;17(20):7552. doi: 10.3390/ijerph17207552. PMID 33080802
- [Background] Debillon T, Zupan V, Ravault N, Magny JF, Dehan M. Development and initial validation of the EDIN scale, a new tool for assessing prolonged pain in preterm infants. Arch Dis Child Fetal Neonatal Ed. 2001 Jul;85(1):F36-41. doi: 10.1136/fn.85.1.f36. PMID 11420320
- [Background] Chooi CS, White AM, Tan SG, Dowling K, Cyna AM. Pain vs comfort scores after Caesarean section: a randomized trial. Br J Anaesth. 2013 May;110(5):780-7. doi: 10.1093/bja/aes517. Epub 2013 Feb 5. PMID 23384734
- [Background] Laksonen RP Jr, Gasiewicz NK. Implementing a Program for Ultrasound-Guided Peripheral Venous Access: Training, Policy and Procedure Development, Protocol Use, Competency, and Skill Tracking. Nurs Clin North Am. 2015 Dec;50(4):771-85. doi: 10.1016/j.cnur.2015.07.010. PMID 26596664
- [Background] Lamperti M, Biasucci DG, Disma N, Pittiruti M, Breschan C, Vailati D, Subert M, Traskaite V, Macas A, Estebe JP, Fuzier R, Boselli E, Hopkins P. European Society of Anaesthesiology guidelines on peri-operative use of ultrasound-guided for vascular access (PERSEUS vascular access). Eur J Anaesthesiol. 2020 May;37(5):344-376. doi: 10.1097/EJA.0000000000001180. PMID 32265391
- [Background] Adhikari S, Schmier C, Marx J. Focused simulation training: emergency department nurses' confidence and comfort level in performing ultrasound-guided vascular access. J Vasc Access. 2015 Nov-Dec;16(6):515-20. doi: 10.5301/jva.5000436. Epub 2015 Jun 20. PMID 26109540
- [Background] van Loon FH, Puijn LA, van Aarle WH, Dierick-van Daele AT, Bouwman AR. Pain upon inserting a peripheral intravenous catheter: Size does not matter. J Vasc Access. 2018 May;19(3):258-265. doi: 10.1177/1129729817747531. Epub 2018 Mar 4. PMID 29772984
- [Background] Moore GF, Audrey S, Barker M, Bond L, Bonell C, Hardeman W, Moore L, O'Cathain A, Tinati T, Wight D, Baird J. Process evaluation of complex interventions: Medical Research Council guidance. BMJ. 2015 Mar 19;350:h1258. doi: 10.1136/bmj.h1258. PMID 25791983
- [Derived] Slosse C, Manneville F, Ricci L, Ostermann A, Klein S, Bouaziz H, Ambroise-Grandjean G. Development and evaluation of an algorithm for peripheral venous catheter placement (ALCOV): protocol for a quasi-experimental study. BMJ Open. 2024 Jun 19;14(6):e078002. doi: 10.1136/bmjopen-2023-078002. PMID 38904139